CLINICAL TRIAL: NCT01441284
Title: Efficacy of Pramipexole Extended Release in the Treatment of Essential Tremor: a Double-blind, Cross-over, Placebo-controlled Multicenter Study
Brief Title: Efficacy of Pramipexole Extended Release in the Treatment of Essential Tremor
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dr. Norbert Kovacs, Associate professor, specialist in neurology and movement disorders, Department of Neurology, University of Pecs
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOK_KA_2011_pramipexole; 34039/KA-OTKA/11-10 (Other: University of Pécs, Faculty of Medicine)
Record Dates: First submitted 2011-09-21; First posted 2011-09-27 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Essential Tremor
Keywords: pramipexole; essential tremor; cross-over
MeSH Terms: conditions — Essential Tremor | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Process 1 (Active Comparator): 10 weeks of pramipexole treatment 2 weeks wash-out period (cross-over) 10 weeks placebo treatment
  Interventions: Drug: pramipexole; Drug: placebo
- Process 2 (Placebo Comparator): 10 weeks of placebo treatment 2 weeks wash-out period (cross-over) 10 weeks pramipexole treatment
  Interventions: Drug: pramipexole; Drug: placebo

INTERVENTIONS:
Drug: pramipexole — pramipexole extended release, 2.1 mg pramipexole base (3.0mg pramipexole salt) once daily
  Other Names: Mirapexin retard
Drug: placebo — placebo

SUMMARY:
Aim of the study is to perform a double-blind, crossover, placebo-controlled multicenter study evaluating the efficacy of pramipexole on essential tremor.

DETAILED DESCRIPTION:
Essential tremor is one of the most common movement disorders with the prevalence of 3-5% among the elderly population. Although its main clinical feature is the bilateral, predominantly postural-kinetic tremor, newer studies suggest that ET is a spectrum of clinical features with both motor and nonmotor elements not homogeneously distributed.

Despite its high occurrence, the pharmacological treatment of ET is limited. Although the mainline drugs, propranolol and primidone, can provide good clinical benefit in a portion of cases, >50% of the patients stop the medication due to inefficacy or side-effects. Hypotension, dizziness, bradycardia, cognitive impairment, fatigue and erectile dysfunction are the most common side-effects contributing to medication discontinuation.

In an open-label pilot study, the investigators previously demonstrated that 2.1 mg/day pramipexole extended-release improved both the severity of tremor (by 52%) and health-related quality of life.

The present study aims to confirm this hypothesis in a double-blind, crossover, placebo-controlled multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ET has to be unambiguous based on the clinical diagnostic criteria.
* Tremor has to be severe enough to produce disability.
* Patients must sign a written informed consent according with the approval of the Regional Ethical Board of University of Pécs

Exclusion Criteria:

* Exclusion criteria are established in accordance to the guidelines of Elble et al3.
* Presence of any medical conditions capable of producing tremor (e.g. hyperthyroidism, drug withdrawal, neuropathy, etc.).
* Except for cogwheel phenomenon, the presence of any abnormal neurological signs (e.g. dystonia, myoclonus, ataxia, parkinsonism, cerebellar or pyramidal signs, etc.)
* Atypical tremor appearance for ET (e.g. isolated vocal-cord tremor, orthostatic tremor, task-specific tremor, etc.)
* Presence or suspicion of psychogenic tremor
* Usage of medication capable of producing tremor (e.g. sympathomimetics, valproate, etc.)
* Concomitant administration of any drugs potentially capable of improving ET (e.g. antiepileptics, beta-receptor blockers).
* Previous neurosurgical treatment (e.g. deep brain stimulation or thalamotomy).
* Presence of serious concomitant disorders capable of interfering with the study (e.g. heart failure, tumorous disorders, etc.)
* Presence of any contraindication for pramipexole treatment (e.g. impulsive control disorder, known hypersensitivity to any components of the tablets, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in tremor severity | 10 weeks of treatment
  Improvement in tremor severity measured by Fahn-Tolosa-Marin Tremor Rating Scale

SECONDARY OUTCOMES:
Improvement in quality of life | 10 weeks of treatment
  Improvement in quality of life assessed by EQ-5D score
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 10 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Kovacs, MD, PhD, Principal Investigator — Associate professor
Locations (2):
- Hungary (2):
  - Department of Neurology, University of Pécs, Pécs, Baranya
  - Kaposi Mór County Hospital, Kaposvár, Somogy County

REFERENCES:
- [Background] Kovács N, Pál E, Késmárky I, Komoly S, Nagy F, Herceg M. Pramipexole for treating essential tremor. Eur J Neurol 2011;18(Suppl 2):482.